CLINICAL TRIAL: NCT00278798
Title: TRAIL-CC: Trachelectomy, Radical Hysterectomy, and Intimate Life After Cervical Cancer Study
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Lori Brotto, Principal Investigator, University of British Columbia
Other Study IDs: C05-0591
Record Dates: First submitted 2006-01-16; First posted 2006-01-18 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Cervical Cancer
Keywords: tracehelectomy; radical hysterectomy
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this study is to compare radical hysterectomy with trachelectomy on outcomes related to intimacy, sexual health, and mood immediately before, 1 month after, and 6 months after surgery.

DETAILED DESCRIPTION:
Improvements in our treatment of these cancers has resulted in an increased focus on quality of life issues. Sexual health is one such important aspect of quality of life that is often disrupted in cervical cancer survivors. However, currently there are no established treatments for such sexual problems, often leaving women and their partners with long-term difficulties that interfere in other aspects of their relationship and lives.

Treatment of cervical cancer involves hysterectomy (i.e. removal of the uterus), and commonly bilateral salpingo-oophorectomy (BSO; i.e. bilateral removal of the ovaries and fallopian tubes). Hysterectomy results in direct physical consequences to sexual function which have been attributed to probable autonomic nerve damage (Butler-Manuel et al., 2000; 2002; Weijmar Schultz et al., 1991). Depending on the extent of disease, hysterectomy may be either simple (i.e. surgical removal of the uterus without excision of adjoining tissue) or radical (i.e. surgical removal of the uterus, the parametria and uterosacral ligaments, the upper portion of the vagina, and the pelvic lymph nodes).

In the last two decades, a new procedure known as trachelectomy, has surfaced to treat early stages of cervical cancer. Unlike radical hysterectomy, the trachelectomy procedure aims to preserve the fertility in young women who wish to have children post cervical cancer and treatment (Plante et al., 2004; 2005). This preservation of fertility in trachelectomy is a result of leaving the patient's uterus intact while removing the cervix, parametrium and upper one third of the vagina. With the uterus intact, the patients are capable of conceiving multiple births post-procedure (Bernardini et al., 2003, Plante et al., 2004; 2005), an option that was not present in the past for women after radical hysterectomy.

The few dozen studies done looking at the outcomes of trachelectomy have mainly focused on medical outcomes such as fertility and cancer cure and recurrence. The findings show there is a 70-72% success rate in women who try to conceive post-trachelectomy (Boss et al., 2005, Plante et al., 2005). If a patient is eligible for a trachelectomy procedure, according to the criteria (Sonoda et al., 2004), recurrence-free survival is excellent at 95% (Plante et al., 2004).

With such improvements in the identification and cure of cervical cancer and the use of fertility-sparing techniques, there has been an increase in the number of young patients in remission, raising a number of quality of life issues. Sexual health is recognized as an integral aspect of quality of life during survivorship and is increasingly receiving research and clinical attention (Juraskova et al., 2003; Wenzel et al., 2002). In the studies done on trachelectomy we find that there are a handful of women who, prior to the operation, wish to conceive a child, but post-operation lose this desire and do not try to conceive (Boss et al., 2005, Plante et al., 2005), but no further studies have been done in this area as to the reasons why. Although the studies have been very beneficial for medical information none of the studies examining the efficacy of trachelectomy have studied the impact on sexual health or quality of life. On the other hand, research on the effects of radical hysterectomy in women with cervical cancer finds approximately half of women experience negative sexual side-effects such as significantly more lubrication difficulties, reduced vaginal length and elasticity, and marked distress (Bergmark et al., 1999). Also distressing to 36% of the women in this group is the absence of genital swelling in more than half of their sexual encounters, despite no changes in sexual frequency or orgasmic experience (Bergmark et al., 1999). When a vaginal photoplethysmograph was used to document changes in genital blood flow (an indirect measure of sexual arousal), women with radical hysterectomy had more impairment in blood flow responses than either a control group or a simple hysterectomy group, suggesting involvement of autonomic nerves (Maas et al., 2002).

Given that women, together with their partners and oncologists, may find themselves in a position of selecting one procedure over another, it seems important to better understand the relative effects of these procedures on intimate life and sexual health. The objective of this study, therefore, is to compare radical hysterectomy with trachelectomy in the effects on intimacy, sexual health, and mood immediately before, 1 month after, and 6 months after surgery.

This study will help to identify patterns and outcomes on these aspects of quality of life in hopes of better informing women of the potential outcomes of their procedures. Cervical cancer and treatment are life-altering events; therefore it is desirable to identify and hopefully reduce any negative psychological and physical sequelae of treatment. We want to ensure that problems related to post-cervical cancer are diminished so that the survivor's quality of life can be maintained at an acceptable level, allowing the patients to continue living a fulfilling life, uninhibited by sexual and emotional distress.

ELIGIBILITY:
Inclusion Criteria:

1. Women who have a diagnosis of cervical cancer
2. Women who are scheduled for either a radical hysterectomy or radical trachelectomy at the British Columbia Cancer Agency - Vancouver Cancer Centre
3. Proficient in English

Exclusion Criteria:

No woman who meets the inclusion criteria will be excluded from participating.

Ages: 19 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women diagnosed with cervical or endometrial cancer
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2006-01; Primary Completion 2011-07 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lori A Brotto, PhD, Principal Investigator — University of British Columbia
Locations (1):
- British Columbia Cancer Agency, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Bergmark K, Avall-Lundqvist E, Dickman PW, Henningsohn L, Steineck G. Vaginal changes and sexuality in women with a history of cervical cancer. N Engl J Med. 1999 May 6;340(18):1383-9. doi: 10.1056/NEJM199905063401802. PMID 10228188
- [Background] Bernardini M, Barrett J, Seaward G, Covens A. Pregnancy outcomes in patients after radical trachelectomy. Am J Obstet Gynecol. 2003 Nov;189(5):1378-82. doi: 10.1067/s0002-9378(03)00776-2. PMID 14634572
- [Background] Boss EA, van Golde RJ, Beerendonk CC, Massuger LF. Pregnancy after radical trachelectomy: a real option? Gynecol Oncol. 2005 Dec;99(3 Suppl 1):S152-6. doi: 10.1016/j.ygyno.2005.07.071. Epub 2005 Sep 2. PMID 16140367
- [Background] Butler-Manuel SA, Buttery LD, A'Hern RP, Polak JM, Barton DP. Pelvic nerve plexus trauma at radical hysterectomy and simple hysterectomy: the nerve content of the uterine supporting ligaments. Cancer. 2000 Aug 15;89(4):834-41. doi: 10.1002/1097-0142(20000815)89:43.0.co;2-7. PMID 10951347
- [Background] Butler-Manuel SA, Buttery LD, A'Hern RP, Polak JM, Barton DP. Pelvic nerve plexus trauma at radical and simple hysterectomy: a quantitative study of nerve types in the uterine supporting ligaments. J Soc Gynecol Investig. 2002 Jan-Feb;9(1):47-56. doi: 10.1016/s1071-5576(01)00145-9. PMID 11839509
- [Background] Juraskova I, Butow P, Robertson R, Sharpe L, McLeod C, Hacker N. Post-treatment sexual adjustment following cervical and endometrial cancer: a qualitative insight. Psychooncology. 2003 Apr-May;12(3):267-79. doi: 10.1002/pon.639. PMID 12673810
- [Background] Plante M, Renaud MC, Francois H, Roy M. Vaginal radical trachelectomy: an oncologically safe fertility-preserving surgery. An updated series of 72 cases and review of the literature. Gynecol Oncol. 2004 Sep;94(3):614-23. doi: 10.1016/j.ygyno.2004.05.032. PMID 15350349
- [Background] Plante M, Renaud MC, Hoskins IA, Roy M. Vaginal radical trachelectomy: a valuable fertility-preserving option in the management of early-stage cervical cancer. A series of 50 pregnancies and review of the literature. Gynecol Oncol. 2005 Jul;98(1):3-10. doi: 10.1016/j.ygyno.2005.04.014. PMID 15936061
- [Background] Sonoda Y, Abu-Rustum NR, Gemignani ML, Chi DS, Brown CL, Poynor EA, Barakat RR. A fertility-sparing alternative to radical hysterectomy: how many patients may be eligible? Gynecol Oncol. 2004 Dec;95(3):534-8. doi: 10.1016/j.ygyno.2004.07.060. PMID 15581959
- [Background] Wenzel LB, Donnelly JP, Fowler JM, Habbal R, Taylor TH, Aziz N, Cella D. Resilience, reflection, and residual stress in ovarian cancer survivorship: a gynecologic oncology group study. Psychooncology. 2002 Mar-Apr;11(2):142-53. doi: 10.1002/pon.567. PMID 11921330
- [Background] Weijmar Schultz, W. C. M., van de Wiel, H. B. M. & Bouma, J. (1991) Psychosexual functioning after treatment for cancer of the cervix: A comparative and longitudinal study. Int J Gynecol Cancer, 1, 37-46.